CLINICAL TRIAL: NCT02839226
Title: Prospective, Placebo-controlled, Double-blind, Randomized Clinical Study to Assess the Safety and Efficacy of Topical Treatment of AR/101 Compared With for up to 28 Days, in Accelerating Granulation Tissue Formation in Chronic Wound Patients
Brief Title: Safety and Efficacy of Topical AR/101 Compared With Placebo, in Accelerating Granulation Tissue Formation of Hard-to-heal Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Arava Bio Tech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-H2H-2016-04
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Wounds; Other Ulcers Wounds and Skin Problems
Keywords: ulcers; wounds; diabetes; venous ulcers; arterial ulcers; granulation tissue; protein kinase c
MeSH Terms: conditions — Wounds and Injuries; Ulcer; Diabetes Mellitus; Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AR/101 (Active Comparator): AR/101 will be administered topically once daily for up to 28 days concomitantly with standard of care as advised by treating physician. After randomization, patients will be treated for up-to 28 days, or until granulation tissue formation has reached maximal score on the granulation scale, or until the wound is ready for skin grafting, whichever occurs first.
  Interventions: Drug: AR/101
- Placebo (Placebo Comparator): placebo will be administered topically once daily for up to 28 days concomitantly with standard of care as advised by treating physician. After randomization, patients will be treated for up-to 14 days or until granulation tissue formation has reached maximal score on the granulation scale, or until the wound is ready for skin grafting, whichever occurs first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR/101
  Arms: AR/101
Drug: Placebo
  Arms: Placebo

SUMMARY:
This prospective, placebo-controlled, double blind, randomized study is designed to assess the healing effects of AR/101 on chronic Hard-to-Heal wound(s) of different etiologies including arterial ulcers, diabetic ulcers and venous ulcers, of at least 3 months duration. After collection of comprehensive medical data to confirm eligibility of patient and obtaining informed consent , patients will enter Screening run-in Period where all wounds will be cleaned if necessary by surgical debridement and irrigation (isotonic solution) prior to initiation (run-in phase) of the study according to physician's instructions. During the 14 day screening period, all subjects will receive standard of care (SoC) on a daily basis, as per indication and patients status, according to physicians instructions. Wounds will be morphologically assessed by the treating physician and by photographic evaluation by the PI once a week - at days 7 and 14 of the screening run-in phase. Following the run-in period, Subjects with wounds of ≥ 5cm2 and ≤100 cm2 of at least 3 months duration that fail to respond to treatment with SoC during the screening run-in phase will be enrolled into the study. Eligible subjects with wounds will be randomized and treated topically with AR/101+ SoC or placebo +SoC once daily for up to 14 days. During this treatment phase I, depending on their wound size and wound type, subjects will receive treatment dose applied topically daily and wounds will be dressed according to physician's instructions. Wounds will be photographed daily and assessed by the treating physician in the clinic once a week (at the end of each weekly period). During the treatment period, adverse events and concomitant medications will be monitored; wounds will be morphologically assessed by photo documentation and followed for wound bed progression and granulation tissue formation. At the end of Treatment period I, patient's wounds will be analyzed and all patients from both treatment arms with wound score 0-2 will be assigned to receive the study drug for and additional up to 14 days treatment phase II in full accordance with the treatment regimen described in Treatment phase I. A termination visit will be performed at day 14 of Treatment phase I or II or earlier if the wound has reached the maximum score on the granulation scale or if the wound is ready for skin grafting; or in any case of early withdrawal that is not due to withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years old and above
2. Have single/multiple wounds
3. Have a chronic hard to heal wound of various etiologies for at least 3 months of duration
4. Patient was treated for 14 days with SoC (screening run-in) and did not respond to treatment. "Response" is defined as formation of more than 10% of viable granulation tissue.
5. Wound area is larger than 5cm2 and smaller than 100 cm2.
6. Subject should be available for the entire study period, and be able and willing to adhere to protocol requirements
7. Subject must sign an informed consent form prior to undergoing any study- related procedures.
8. For female subjects only, the subject is either:

A. Surgically sterile B. At least 1 year post-menopausal.

C. Subject has consented to using one of the following acceptable methods of birth control for the times specified below:

* Intra-uterine device (IUD) in place for at least 3 months prior to screening visit and through study completion.
* Barrier method (condom or diaphragm) for at least 14 days prior to screening through study completion.
* Spermicide for at least 14 days prior to screening through study completion.
* Stable hormonal contraceptive for at least 3 months prior to screening visit through study completion.
* Surgical Sterilization (vasectomy) of partner at least 6 months prior to screening visit through study completion.

Exclusion Criteria:

1. Have a documented medical history of a significant hematological, cardiac, pulmonary, gastrointestinal, endocrine (other than Diabetes Mellitus type 1 or 2), or hepatic disease which per the physician's discretion prohibit them from entering the study.
2. Had any clinically significant illness per the physician's discretion during the last 4 weeks prior to the screening period.
3. Have a documented medical history . of HBV, HCV, HIV.
4. Severely immunosuppressed for any reason that would limit or preclude healing in the opinion of the Investigator.
5. Patient is currently receiving, or has received at any time within one month prior to enrollment, any medications or treatments known to affect the wound healing processes including Glucocorticosteroid treatment (Prednisone > 10mg/day or its equivalent), immuno-suppressive drugs, radiation therapy and chemotherapy.
6. Use of growth factors, allogeneic skin grafts/ skin graft products within one month prior to enrollment.
7. Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 1 year and not using a medically approved method of contraception (i.e., oral, transdermal, or implanted contraceptives, intrauterine device, diaphragm, condom, abstinence, or surgical sterility), or females who test positive on a blood-based pregnancy test.
8. Clinically significant blood and urinalysis tests per the physician's discretion.
9. Have any acute signs of infection in the wound, which could be linked to raised body temperature, abscess, necrosis, cellulitis or acute osteomyelitis.
10. Have sinus tracts or tunnels, purulent discharge , gangrene or severe drainage that will cause skin maceration per the physician's discretion.
11. Had any antibiotic treatment for acute infection during the screening period (prophylactic antibiotic treatment is allowed)
12. Intolerance to compression therapy if required for venous ulcers or inability to follow SoC according to the physician's instructions.
13. Had revascularization surgery during the past 3 months or be a candidate for revascularization surgery during the course of the study.
14. Active wound care therapies within the past 3 months (e.g., manufactured dermis, full-thickness skin, Becaplermin, split thickness autologous skin grafts at the site of the target wound)
15. Patients with poor nutritional status (albumin < 2.5g/dl), poor diabetic control (HbA1c > 12%), anemia (hemoglobin<8 g/dL), a leukocyte counts < 4,000// μl or >15000/μl, renal failure (Cr > 3 mg/dl);
16. Active deep venous thrombosis (DVT)
17. Patients with uncontrollable edema >+2
18. Patients who in the opinion of the investigator, for any reason other than those listed above will not be able to complete the study per protocol.
19. Participation in another clinical trial within 30 days prior to the Screening period or during this study.
20. History of mental illness that would preclude completion of the study

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
comparison of the formation of new granulation tissue according to a Granulation Score, between the AR/101 treated group and the placebo group, during the treatment phases | 28 days

SECONDARY OUTCOMES:
Percentage of patients ready for skin grafting or healing by secondary intention during treatment phase 1 and treatment phase 2 based on physician's assessment | 28 days
Percent of patient responders of equal or more then 75% granulation tissue during two weeks of treatment phase 1 | 14 days
Mean time to response (equal or more then 75% of granulation tissue) during two weeks of treatment phase 1 | 14 days
Mean time to response (equal or more then 75% of granulation tissue) during two weeks of treatment phase 2 | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel